CLINICAL TRIAL: NCT05229731
Title: Description of the Neurovisual and Radiological Specificities of Patients With Visual Snow
Brief Title: Description of the Neurovisual and Radiological Specificities of Patients With Visual Snow Syndrome
Acronym: NEVICOG
Status: Withdrawn | Type: Observational
Why Stopped: The investigators no longer want to do the project
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NDO_2021_17
Record Dates: First submitted 2021-09-10; First posted 2022-02-08 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Visual Snow Syndrome
Keywords: Visual Snow Syndrome
MeSH Terms: conditions — visual snow syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients with visual snow syndrome according to international criteria
  Interventions: Procedure: Neurovisual evaluation; Procedure: Cerebral MRI
- Control group: Patients without visual snow syndrome according to international criteria
  Interventions: Procedure: Neurovisual evaluation; Procedure: Cerebral MRI

INTERVENTIONS:
Procedure: Neurovisual evaluation — Standardized tests and scales classically used during a neurovisual evaluation,
Procedure: Cerebral MRI — Sequences realized :
  * 3D T1 TFE i1.0
  * 3D FLAIR i1.0
  * 2D T2 0.3 coro, centré sur les orbites
  * 3D T2 i0.6
  * SWIp 0.6
  * 3D PD T2 NO, centré sur les orbites
  * 3D ASL
  * DTI 64dir

SUMMARY:
NEVICOG is a single-center study evaluating neurovisual and radiological specificities in patients with visual snow syndrome (VSS) compared to a control population.

DETAILED DESCRIPTION:
Visual snow syndrome (SNV) is characterized by a continuous grainy or pixelated visual sensation additional to the perceived image. Patients often report a feeling similar to seeing noise from cathode-ray televisions.

The prevalence is not well known but about 2% of the population could be reached. Although benign and stable, this pathology is often troublesome in everyday life.

Its precise etiology remains unknown to this day. Ophthalmologic explorations do not reveal any significant abnormalities. Neurologically, "standard" examinations appear normal. Only the examinations carried out in the context of research have been able to highlight anomalies such as an imbalance between visual cortical inhibition and excitation as well as a high spontaneous neural triggering and hypermetabolism of the associative visual cortex (functional MRI, PET- MRI). In addition, the Visual Evoked Potentials show a lack of habituation, testifying to cortical hyperexcitability.

To our knowledge, no specific neurovisual study focusing on the functions involved in the processing of visual information has been carried out to date. We propose the realization of a complete evaluation made up of existing tasks as well as the adaptation of some of them specific to SNV.

The posterior abnormalities currently highlighted by imaging have been carried out in examinations not available on a daily basis. A non-invasive brain MRI study will be carried out in our patients using more recent techniques (MRI with arterial spin labelling or ASL for Arterial Spin Labelling, and diffusion tensor imaging or DTI for Diffusion Tensor Imaging) in order to search for possible posterior lesions and clinical radiological correlations.

Thus, this study aims to carry out a more in-depth neurovisual exploration of this syndrome, in order to allow a better understanding of this frequent and disabling disorder on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

Case group:

* Patient aged up to 55
* Diagnosis of visual snow syndrome according to the international criteria
* Visual snow symptoms still present
* Express consent to participate in the study

Control group:

* Person aged up to 60
* Matched to an SNV patient on age (+/- 5 years) and sex
* Express consent to participate in the study

Exclusion Criteria:

Case group:

* Patient with an absolute or relative contraindication to MRI (claustrophobia, incompatible implantable device, etc.)
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* Non-French speaking patient
* Added psychiatric or neurodegenerative pathology unrelated to visual snow likely to induce neurocognitive and neurovisual disorders in the short or long term
* Ophthalmologic comorbidity that may interfere with the interpretation of examinations

Control group:

* Patient with an absolute or relative contraindication to MRI (claustrophobia, incompatible implantable device, etc.)
* Person benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* Non-French speaking person
* Psychiatric or neurodegenerative pathology likely to induce neurocognitive and neurovisual disorders in the short or long term
* Ophthalmologic comorbidity that may interfere with the interpretation of examinations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with of visual snow syndrome according to international criteria compared to control patients without any visual snow syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04-13 (Estimated); Primary Completion 2022-04-13 (Estimated); Study Completion 2022-04-13 (Estimated)

PRIMARY OUTCOMES:
Results of the neurovisual assessment | 1 day (Inclusion)
  Rey-Osterrieth test will be used to assess the neurovisual ability. Patients have to reproduce a figure composed of 18 elements. A score between 0 and 2 is given to each of these elements according to their accuracy. The score varies from 0 to 36 and assesses the patient's visuo-constructive ability (36 corresponds to the best visuo-constructive ability).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Di Donato, Principal Investigator — Hôpital Fondation A. de Rothschild; Romain Deschamps, MD, Study Director — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France